CLINICAL TRIAL: NCT02235545
Title: Optisure Lead Post Approval Study
Status: Terminated | Type: Observational
Why Stopped: Abbott received FDA approval to transition the ongoing Optisure PAS to a Real World Evidence methodology through the EP Passion project
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 60045220
Record Dates: First submitted 2014-09-07; First posted 2014-09-10 (Estimated); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Tachycardia, Ventricular
Keywords: High Voltage (HV) Lead; Implantable Cardioverter Defibrillator (ICD); cardiac resynchronization therapy defibrillator (CRT-D) System; Treatment of Heart Failure; Treamtent of life-threatening ventricular tachyarrhythmia; Optisure
MeSH Terms: conditions — Heart Failure; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- St. Jude Medical Optisure Lead: Patients implanted with St. Jude Medical Optisure Lead
  Interventions: Device: St. Jude Medical Optisure Lead

INTERVENTIONS:
Device: St. Jude Medical Optisure Lead — Patients implanted with St. Jude Medical Optisure Lead

SUMMARY:
The purpose of this post approval study is to characterize the chronic performance of the SJM Optisure family of HV leads in patients.

DETAILED DESCRIPTION:
The Optisure lead study is a multi-center, post-approval study that will be performed in compliance with the Conditions for Approval, as agreed upon with the FDA. Patients will be permitted to enroll in the study up to 30 days post-implant of the Optisure lead. Following a successful implant, patients will be followed every 6 months until 60 months (5 years). After patients complete 60 months of follow-up, their participation in the study will end. Patients who are consented prior to implant and for whom an implant is unsuccessful will be followed for 30 days for any adverse events and then withdrawn from the study, or may have an implant reattempted if the physician and patient choose to do so.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will meet all of the following:

1. Have an approved indication, as per ACC/AHA/HRS/ESC guidelines, for implantation of an ICD or CRT-D system for treatment of heart failure or life-threatening ventricular tachyarrhythmia(s).
2. Have been implanted with a St. Jude Medical Optisure lead in the last 30 days or are scheduled for an Optisure lead implant.
3. Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations.
4. Are 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

Patients will be excluded if they meet any of the following:

1. Enrolled or intend to participate in a clinical drug and/or device study, which could confound the results of this trial as determined by SJM, during the course of this clinical study.
2. Have a life expectancy of less than 5 years due to any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD/CRT-D indicated patients
Sampling Method: Non-Probability Sample
Enrollment: 1735 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (60):
- United States (46):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - St. Bernards (formerly Cardiology Associates of Northeast Arkansas), Jonesboro, Arkansas
  - Raymond Schaerf, MD, Burbank, California
  - Desert Heart Rhythm Consultants, Palm Springs, California
  - Cardiac Rhythm Specialists, Inc., Reseda, California
  - San Diego Heart Rhythm Center (formerly San Diego Heart and Vascular Associates), San Diego, California
  - Jorge Diaz, M.D. , P.A., Lake Mary, Florida
  - Northside Hospital, Atlanta, Georgia
  - Rockford Cardiology Associates, Rockford, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - St. Elizabeth Medical Center - South Unit, Edgewood, Kentucky
  - Peninsula Cardiology Associates, Salisbury, Maryland
  - Mass Heart & Rhythm, Leominster, Massachusetts
  - Premier Medical Clinics, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Northern Michigan Hospital, Traverse City, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - HealthCare Partners Cardiology, Las Vegas, Nevada
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Cardiovascular Group of Syracuse, Liverpool, New York
  - High Point Regional Health (formerly Carolina Cardiology Cornerstone), High Point, North Carolina
  - CarolinaEast Heart Center, New Bern, North Carolina
  - VA Medical Center Cleveland, Cleveland, Ohio
  - Great Lakes Medical Research, LLC, Willoughby, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Arrhythmia Institute, Newtown, Pennsylvania
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - HeartPlace, Bedford, Texas
  - VA Medical Center Dallas, Dallas, Texas
  - Cardiology Care Consultants, El Paso, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Heart of Dixie Cardiology (formerly Dixie Regional Medical Center - River Road Campus), St. George, Utah
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Aurora Medical Group, Milwaukee, Wisconsin
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium
- Canada (7):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - QE II Health Sciences, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Rouge Valley Centenary, Scarborough Village, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
- Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Germany
- Japan (3):
  - Tokyo Women's Medical University, Shinjuku-Ku, Kanto
  - Osaka City University Hospital, Abeno-ku, Osaka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
- Mc-Tronik, Lodz, Poland
- Santa Maria Hospital, Lisbon, Lisbon District, Portugal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | St. Jude Medical Optisure Lead
Started | 1735 (Total Subject Cohort)
Withdrawal Before 12 Month (12M) Follow-up (FU) Visit | 102
Deaths Before 12M FU Visit | 101
Completed 12M FU Visit | 1389
Withdrawals Before 24M FU Visit | 107
Deaths Before 24M FU Visit | 89
Completed 24M FU Visit | 1203
Withdrawals Before 36M FU Visit | 93
Deaths Before 36M FU Visit | 70
Completed 36M FU Visit | 1023
Withdrawals Before 48M FU Visit | 55
Deaths Before 48M FU Visit | 56
Completed 48M FU Visit | 483
Withdrawals Before 60M FU Visit | 11
Deaths Before 60M FU Visit | 7
Completed (60 FU Visit) | 14
Not Completed | 1721

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: Patients implanted with St. Jude Medical Optisure Lead
  St. Jude Medical Optisure Lead: Patients implanted with St. Jude Medical Optisure Lead
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 1735
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 399
  Male | 1336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 106
  Not Hispanic or Latino | 1568
  Unknown or Not Reported | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9
  Asian | 53
  Black or African American | 188
  Native Hawaiian or Other Pacific Islander | 3
  Other | 14
  White | 1409
  Unknown | 59
NYHA Class per Blinded Assessor at Baseline, n(%) [Count of Participants; unit: Participants] — Class I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  Class III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    Class I | 179
    Class II | 712
    Class III | 771
    Class IV | 15
    Not Available | 58
Arrhythmia History, n(%) [Count of Participants; unit: Participants]
  Ventricular Arrhythmias | 564
  Atrial Arrhythmias | 575
Primary CRT-D Indication for Implant, n(%) [Count of Participants; unit: Participants]
  Cardiac Arrest | 91
  CRT - Other | 9
  CRT Generator Change | 8
  Familial Condition | 19
  Heart Failure with Atrial Fibrillation | 59
  Heart Failure with Wide QRS | 379
  ICD - Other | 38
  ICD Generator Change | 13
  Ischemic Cardiomyopathy | 551
  Non-Ischemic Cardiomyopathy | 330
  Reduced ejection fraction with Frequent Dependence on V-Pacing | 49
  Syncope | 29
  Ventricular Tachycardia | 160

OUTCOME MEASURES:

1. Primary Outcome: Complication Free Survival Rate at 5 Years for Complications Related to the Optisure RV Leads.
Description: Freedom from right ventricle (RV) lead related complications within 30 days of implant at 5 years follow-up
  Due to early termination of study, the sample size at 5 years follow-up was insufficient to perform the pre-specified primary endpoint analysis. The endpoint was evaluated using the Kaplan-Meier method however the hypothesis test was not performed due to insufficient sample size. The percentage freedom from RV lead related complications was summarized through 5-years from attempted RV lead implant. For subjects who experienced RV lead related complication, the time to event will be calculated from the attempted implant to the date that the first event occurred. For subjects that did not experience the complication, the time to event was censored at their last known event-free time point.
Time Frame: 5 years
Population: Subjects with an attempted implant.
Measure: Number (95% Confidence Interval); unit: % pts free from RV related complications
Groups:
- St. Jude Medical Optisure Lead: Patients with attempted St. Jude Medical Optisure Lead implanted
Arm/Group | St. Jude Medical Optisure Lead
Number analyzed (Participants) | 1735
% pts free from RV related complications | 96.3 [94.0 to 97.8]

ADVERSE EVENTS:
Time Frame: Up to 5 years from baseline for each participant
Groups:
- Right Ventricle Lead-Related Complications: Summary of RV Lead-Related Complications. A complication is an adverse event caused by or associated with the study device, system component(s), and or procedure that requires invasive intervention (e.g. lead dislodgement requiring repositioning) including RV lead perforations. All RV lead perforations will be reported as complications.
- Summary of System and/or Procedure Related Complications Not Related to the RV Lead.: Summary of System and/or Procedure Related Complications not related to the RV lead. Includes both System/Pule Generator/Lead Related (RA/LV) and Procedure Related Only
Arm/Group | Right Ventricle Lead-Related Complications | Summary of System and/or Procedure Related Complications Not Related to the RV Lead.
All-Cause Mortality (participants affected / at risk) | 323/1735 | 323/1735
Serious Adverse Events (participants affected / at risk) | 58/1735 | 134/1735
Other Adverse Events (participants affected / at risk) | 58/1735 | 137/1735
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Right Ventricle Lead-Related Complications (N=1735) | Summary of System and/or Procedure Related Complications Not Related to the RV Lead. (N=1735)
Cardiac Perforation (Surgical and medical procedures) | 4 (4) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Elevated Pacing Thresholds (Cardiac disorders) | 7 (7) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 40 (40)
Lead Dislodgement or Migration (Product Issues) | 37 (38) | 40 (48)
Lead Fracture (Product Issues) | 1 (1) | 0 (0)
Lead Noise (Product Issues) | 1 (1) | 1 (1)
Loss of Capture (Product Issues) | 2 (2) | 2 (2)
Oversensing (Product Issues) | 2 (2) | 0 (0)
Pericardial Effusion (Product Issues) | 1 (1) | 1 (1)
Twiddler's Syndrome (Cardiac disorders) | 2 (2) | 3 (3)
Undersensing (Product Issues) | 1 (1) | 0 (0)
Other (Product Issues) | 3 (3) | 3 (3) — One (1) unsuccessful DFT test, resulting in implanting a new lead, one (1) loose suture sleeve, and one (1) lead malfunction
Abnormal Lead Pacing Impedance (Product Issues) | 0 (0) | 1 (1)
Acceleration of Arrhythmias (Product Issues) | 0 (0) | 1 (1)
Device Migration (Surgical and medical procedures) | 0 (0) | 1 (1)
Erosion (Product Issues) | 0 (0) | 3 (3)
Generator Malfunction (Product Issues) | 0 (0) | 10 (10)
Inappropriate Delivery of Therapy (Product Issues) | 0 (0) | 5 (5)
Lead/Port Damage (Product Issues) | 0 (0) | 2 (2)
Phrenic Nerve / Diaphragmatic Stimulation (Product Issues) | 0 (0) | 6 (6)
Thromboemboli (Product Issues) | 0 (0) | 5 (5)
Atrial Arrhythmia (Surgical and medical procedures) | 0 (0) | 1 (1)
Dressler's Syndrome (Surgical and medical procedures) | 0 (0) | 1 (1)
Exacerbation of Heart Failure (Surgical and medical procedures) | 0 (0) | 1 (1)
Formation of Hematomas or Cysts (Surgical and medical procedures) | 0 (0) | 8 (8)
Hemothorax (Surgical and medical procedures) | 0 (0) | 1 (1)
ICD Site Discomfort (Surgical and medical procedures) | 0 (0) | 1 (1)
Pericardial Effusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Pneumothorax (Surgical and medical procedures) | 0 (0) | 3 (3)
Ventricular Arrhythmia (Surgical and medical procedures) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Right Ventricle Lead-Related Complications (N=1735) | Summary of System and/or Procedure Related Complications Not Related to the RV Lead. (N=1735)
Abnormal Lead Defibrillation Impedance <=20 ohms or >=100 ohms (Product Issues) | 1 (1) | 1 (1)
Abnormal Lead Pacing Impedance <=200 ohms or >=200 ohms (Product Issues) | 1 (1) | 1 (2)
Elevated Pacing Thresholds (Product Issues) | 9 (10) | 13 (13)
Inappropriate Delivery of Therapy (Product Issues) | 5 (5) | 28 (32)
Lead Dislodgement or Migration (Product Issues) | 1 (1) | 3 (3)
Lead Noise (Product Issues) | 8 (8) | 10 (12)
Loss of Capture (Product Issues) | 1 (1) | 5 (5)
Oversensing (Product Issues) | 33 (36) | 16 (17)
Phrenic Nerve / Diaphragmatic Stimulation (Product Issues) | 1 (1) | 14 (17)
Other (Product Issues) | 2 (2) | 5 (5) — RV-related: 1 shortness of breath due to RV pacing and 1 lead malfunction (unresolved as of March 2020) Non-RV-lead: 1 chest discomfort, 1 case fatigue and shortness of breath, 1 unsuccessful ATP therapy, 1 generator migration, 1 itching at site
Allergic reaction (Product Issues) | 0 (0) | 3 (3)
Back-Up Device Operation (Product Issues) | 0 (0) | 3 (3)
Failure to Detect VT/VF (Product Issues) | 0 (0) | 4 (4)
Fatigue (Due to Device Programming) (Product Issues) | 0 (0) | 1 (1)
Infection (Surgical and medical procedures) | 0 (0) | 8 (8)
Pacemaker Mediated Tachycardia (PMT) (Product Issues) | 0 (0) | 3 (3)
Pectoral Stimulation (Product Issues) | 0 (0) | 5 (5)
Undersensing (Product Issues) | 0 (0) | 3 (3)
Bleeding (Surgical and medical procedures) | 0 (0) | 3 (3)
Deep Vein Thrombosis (Surgical and medical procedures) | 0 (0) | 2 (2)
Formation of Hematomas or Cysts (Surgical and medical procedures) | 0 (0) | 25 (25)
ICD Site Discomfort (Surgical and medical procedures) | 0 (0) | 1 (1)
Pericardial Effusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Suture Abscess (Surgical and medical procedures) | 0 (0) | 1 (1)
Thromboemboli (Surgical and medical procedures) | 0 (0) | 4 (4)
Ventricular Arrhythmia (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-12-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT02235545/Prot_000.pdf